CLINICAL TRIAL: NCT06579040
Title: The HEROES Trial: Hyperbaric Oxygen Therapy for Endometriosis-Related Pain: A Prospective Randomized Study
Brief Title: The HEROES Trial: Hyperbaric Oxygen Therapy for Endometriosis-Related Pain
Acronym: HEROES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6201
Record Dates: First submitted 2024-08-09; First posted 2024-08-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis-related Pain
Keywords: Endometriosis; Endometriosis-related Pain; Hyperbaric Oxygen Therapy; HBOT
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All possible steps will be taken to maintain blinding of the patient's treating physician (i.e., gynecologist) and assessors. The gynecologist will be blinded to the patient's randomization and patients will be instructed not to disclose their allocated group to their gynecologist and/or research assistants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Control) (No Intervention): Standard multi-modal therapy
- Group II (Intervention) (Experimental): Standard multi-modal therapy + 40 HBOT treatments (2 ATM for 90 mins daily, 5 days a week)
  Interventions: Device: Monoplace Hyperbaric Chamber (Class III medical device)

INTERVENTIONS:
Device: Monoplace Hyperbaric Chamber (Class III medical device) — Participants in the intervention group will be triaged to the closest hyperbaric facility to their address and treated with 40 HBOTs (2 ATM for 90 mins, scheduled daily from Monday to Friday). As HBOT is not a service currently offered at Sunnybrook Hospital, all HBOT treatments will be provided at three collaborating outpatient facilities, Halton Hyperbaric Unit, Restore Hyperbaric Oxygen & Medical Centre (CPSO-certified Level-II OHP), and Rouge Valley Hyperbaric Medical Centre. All three facilities have the exact same hyperbaric chambers, run by anesthesiologists with advanced training, thus treatments will be identical at all sites.
  Arms: Group II (Intervention)

SUMMARY:
Endometriosis, is a condition where tissue from the uterus, called endometrium, grows outside of the uterus. This effects up to 10% of women, and can lead to long-lasting, moderate to severe pelvic pain, infertility and other symptoms. This can affect a woman's quality of life (including increased risk of depression and anxiety) and is associated with increased healthcare costs.

Current treatments are often limited by serious side effects, and many women resort to surgery. Surgery is also associated with complications and there are long wait times for procedures, sometimes over 3 years. This means that many women continue to suffer from symptoms while they wait for surgery. Therefore, new effective treatments for endometriosis pain are needed.

New research suggests that inflammation and stress caused by lack of oxygen in the affected areas may cause endometriosis. Hyperbaric Oxygen Therapy (HBOT), where patients are placed in a small chamber with higher than normal levels of oxygen, suppresses inflammation and promotes tissue healing. Because inflammation is central to this condition, HBOT has emerged as a potential treatment.

In this study, the investigators will test if HBOT, in addition to the standard treatments, is more effective at treating endometriosis pain than the standard treatments alone.

DETAILED DESCRIPTION:
Endometriosis is caused when endometrial-like tissue is found outside of the uterus. It predominantly affects women of reproductive age, with an estimated prevalence of 10% worldwide. Chronic pain related to endometriosis is one of the primary manifestations that lead individuals to seek treatment, with many women reporting moderate to severe pain that can have serious consequences for mental health and quality of life.

Current therapeutic approaches for endometriosis include hormonal therapies (e.g. oral contraceptive pills, progestins, and Gonadotropin-Releasing Hormone agonists/antagonists). While these treatments may provide temporary symptom relief, they are often associated with serious side effects and preclude conception during treatment. The efficacy of other medical interventions remains controversial, therefore surgical procedures are often indicated. However, surgery also has associated risks, has long wait times (between 6 months and 3 years), and a considerable percentage of patients experience recurrence of pain following surgical resection.

Pathologically, endometriosis is characterized by angiogenesis, inflammation, and a chronic hypoxic state at the cellular level. Because of this, Hyperbaric Oxygen Therapy (HBOT), which suppresses inflammation and promotes tissue healing, offers promise as a novel therapeutic modality. This is supported by murine models, which demonstrate the ability of HBOT to reduce inflammation and inflammatory cytokines in the context of endometriosis in animals. However, there have not been any human studies investigating the use of HBOT for treatment of endometriosis and related pain.

This study aims to explore HBOT as a treatment for endometriosis related pelvic pain. Specifically, the investigators will test if HBOT, in addition to the standard treatments (e.g. hormonal and non-hormonal medical options), is more effective at treating endometriosis pain than the standard treatments alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients having refractory pelvic pain (NRS≥4) secondary to endometriosis for >6 months
* May or may not be on traditional multi-modal treatment (pharmacological and/or non-pharmacological)
* On waitlist for surgical treatment

Exclusion Criteria:

* Patients with chronic pain resulting from disease processes unrelated to the pathophysiology of endometriosis-related symptoms (e.g. irritable bowel syndrome, migraine headache, fibromyalgia, chronic low back pain, and musculoskeletal injuries)
* Contraindications/medically unfit to receive hyperbaric treatments at an outpatient facility (e.g. pneumothorax, in-patients, requiring infusions to maintain hemodynamics, active and unstable coronary disease)
* Unlikely to comply with follow-up assessments (e.g. no fixed address, plans to move out of town)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain symptoms on the NRS | At baseline, weekly for the first 8 weeks after enrollment, then at 3/4/5/6 month follow ups
  Assessed on the numeric rating scale between 0 to 10, with 10 indicating the worst possible pain

SECONDARY OUTCOMES:
Change in opioid consumption | At baseline, weekly for the first 8 weeks after enrollment, then at 3/4/5/6 months
  Collected as a categorical variable ("Are you taking 1) more, 2) same or 3) less compared to start of treatment?")
Participant Quality of Life on the EHP-30 | At baseline, and every month for 6 months
  The Endometriosis Health Profile-30 is a validated, high-sensitivity, 30-item endometriosis-specific assessment tool for capturing the impact of endometriosis on patient's lives.
Participant Quality of Life on the SF-36 | At baseline, and every month for 6 months
  The Quality of Life Short Form Survey-36 is a widely used tool to assess an individual's overall health-related quality of life.

OTHER OUTCOMES:
Adherence to HBOT protocol | At 8 weeks (or last session)
  How many patients complete protocol (minimum 4 treatments per week with >35 treatments)
Satisfaction assessed by a Patient Satisfaction Questionnaire | At 8 weeks (or last session) and 6 months following enrollment
  Subjective questionnaire completion at end of treatment inquiring about HBOT experience, barriers to and promoters of treatment
Cost of study completion | Throughout study completion, an average of 6 months
  Cost of study completion on a per patient basis including research support, healthcare resource costs, and patient-related personal costs (transport, time from work)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available following publication of the full trial results.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.